CLINICAL TRIAL: NCT02110927
Title: Microcurrent and Aerobic Exercise Effects in Glycerol, Catecholamines, Energetic Source and Muscle Activity
Brief Title: Microcurrent and Aerobic Exercise Effects in Abdominal Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Andreia Noites, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AN-003
Record Dates: First submitted 2014-03-21; First posted 2014-04-10 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Obesity, Abdominal
Keywords: Abdominal fat; Metabolic syndrome; Microcurrent; Aerobic exercise; Lipolysis
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcutaneous microcurrent (Experimental): This group performed aerobic exercise just after microcurrent in the abdominal region with four transcutaneous electrodes in a parallel position, intensity below the sensitivity threshold and a maximum of 1 milliampere (mA). Every 20 minutes changed from 25 hertz (Hz) to 10 Hz
  Interventions: Device: Transcutaneous microcurrent; Device: Aerobic exercise
- Control group (Placebo Comparator): Control group performed aerobic exercise just after microcurrent in the abdominal region with four transcutaneous electrodes in a parallel position, but microcurrent device was switched off.
  Interventions: Device: Aerobic exercise

INTERVENTIONS:
Device: Transcutaneous microcurrent — Microcurrent in the abdominal region with four transcutaneous electrodes in a parallel position, intensity below the sensitivity threshold and a maximum of 1 mA. Every 15 minutes changed from 25 Hz to 10 Hz.
  Arms: Transcutaneous microcurrent
Device: Aerobic exercise — 50 minutes of aerobic moderate-intensity exercise (45-55% of maximal oxygen consumption (VO2 max)) using Karvonen´s formula, performed on a cycloergometer. Were used Borg scale (12-13), Polar® heart monitors to control heart rate and K4b2 to analyze the quantity of oxygen (O2) consumption and carbon dioxide (CO2) produced during exercise.

SUMMARY:
The purpose of this study was to analyze microcurrent short term effects used with aerobic exercise on abdominal fat.

DETAILED DESCRIPTION:
Nutritional patterns have been changed during twenty-first century with sugar and fat's high proportions that allied to sedentary lifestyle increased body fat. There is already a well establish relationship between total body fat excess, cardiometabolic diseases and increased mortality, knowing that abdominal fat (android pattern), different from body index, presents an additional influence to health risks. Women with their abdominal adipocytes (visceral fat) show an increased lipolytic activity that releases free fat acids to the systemic and portal circulation leading to a metabolic syndrome, increasing the risk of cardiovascular diseases.

Aerobic exercise is a way to decrease fat as it stimulates lipolysis through an increase in catecholamine's level resulting from a sympathetic system nervous activity raise. The most used exercise for lipid elimination is the prolonged aerobic moderate exercise with a minimum of 30 minutes.

Nevertheless aerobic exercise practice reduce globally lipidic sources and not locally .

Electrolipolysis using microcurrent has been used in clinical practice as a technique to reduce abdominal fat. This technique can be applied transcutaneously or percutaneously seeming that the former is not so effective as skin can be an obstacle to the current effect on visceral and subcutaneous fat .

Abdominal fat excess is associated with cardiometabolic diseases and can be prevented using microcurrent and aerobic exercise to stimulate lipolysis.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 30 years.

Exclusion Criteria:

* submitted to other fat reduce procedure, to show cardiovascular risk factors or diseases and/or any physical condition limiting aerobic exercise. To present any contraindications to microcurrent and/or aerobic exercise, to take medication that influence lipid metabolism, and to be pregnant.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in catecholamines and glycerol concentrations | 10 minutes before the interventions, after interventions (duration of interventions - 90 minutes) and after 24 hours
  Blood analysis collection was carried out with help from an clinical analysis technician. The volunteers were not fasting.
Change in proportion of energy source | Immediately before (for 3 minutes) and during exercise (duration of exercise - 50 minutes)
  K4b2 (COSMED ®) was used for analysis of cardiopulmonary gas exchange in real time.
Change in electromyographic activity | 5 minutes before and after microcurrent
  Recording the surface electrical activity produced by rectus abdominis and external oblique in front bridge and side bridge exercise, respectively.

SECONDARY OUTCOMES:
Subcutaneous abdominal fat and visceral abdominal fat | 20 minutes before the interventions
  Ultrasound was performed at the end of expiration to measure subcutaneous abdominal fat between xiphoid apophysis and navel, below navel, and above left and right anterior superior iliac spine. Between xiphoid apophysis and navel was also measured visceral abdominal fat. Abdominal fat analyzed by dual-energy x-ray absorptiometry (DEXA).
Suprailiac, vertical and horizontal abdominal skinfolds | 20 minutes before the interventions
  Suprailiac, vertical and horizontal abdominal skinfolds were performed two times in right hemi body, by caliper.
Perimeters measurements | 20 minutes before the interventions
  The perimeters measurements were done, at the end of expiration, at waist level (below last rib), at navel level, at the point immediately above the iliac crests and at trochanters level. The waist-hip ratio was calculated using the waist level perimeter.
  divided by trochanters level perimeter.
Change in cholesterol, triglycerides and glucose concentrations | 10 minutes before the interventions, after interventions (duration of interventions - 90 minutes)
  Blood analysis collection was carried out with help from an clinical analysis technician. The volunteers were not fasting.

OTHER OUTCOMES:
International Physical Activity Questionnaire | 30 minutes before the interventions
  Used to evaluate the level of physical activity of the volunteers
Food Frequency Questionnaire | 30 minutes before the interventions
  Used to evaluate the lifestyle of the volunteers
Bioimpedance values | 30 minutes before the interventions
  The height was measured with the volunteers on respiratory apnea. To minimize the influence of electrolyte balance changes in bioimpedance assessment, was given some rules to volunteers. It was calculated BMI using the body weight divided by height squared

CONTACTS AND LOCATIONS:
Overall Officials: Andreia Noites, MSc, Principal Investigator — Escola Superior de Tecnologia da Saúde do Porto; Rui Vilarinho, BSc, Study Chair — Escola Superior de Tecnologia da Saúde do Porto
Locations (1):
- Andreia Noites, Vila Nova de Gaia, Porto District, Portugal

REFERENCES:
- [Background] Ahmadian M, Wang Y, Sul HS. Lipolysis in adipocytes. Int J Biochem Cell Biol. 2010 May;42(5):555-9. doi: 10.1016/j.biocel.2009.12.009. Epub 2009 Dec 16. PMID 20025992
- [Background] Despres JP, Lemieux I. Abdominal obesity and metabolic syndrome. Nature. 2006 Dec 14;444(7121):881-7. doi: 10.1038/nature05488. PMID 17167477
- [Background] Bulow J, Gjeraa K, Enevoldsen LH, Simonsen L. Lipid mobilization from human abdominal, subcutaneous adipose tissue is independent of sex during steady-state exercise. Clin Physiol Funct Imaging. 2006 Jul;26(4):205-11. doi: 10.1111/j.1475-097X.2006.00664.x. PMID 16836692